CLINICAL TRIAL: NCT07282496
Title: Evaluation of VEDAN RT-90 Resistant Cassava Starch for Glycemic Control and Prebiotic Fiber Development in a Human Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CS2-25120
Record Dates: First submitted 2025-11-21; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Resistant Starch; Tapioca Starch; Prebiotic Fiber; Blood Sugar
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The first phase of the study was cross-sectional; the second phase was parallel
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RT-90 resistant tapioca starch (Experimental): Phase 1： Equivalent to 50 g total carbohydrates (57 g total product weight) of resistant starch dissolved in 250 mL of water Phase 2： The dosage is calculated at 0.5 grams per kilogram of adult body weight (e.g., a 60-kilogram adult would need to take 30 grams). Subjects should dissolve the test product in water and drink it on an empty stomach before their first meal of the day.
  Interventions: Dietary Supplement: RT-90 resistant tapioca starch
- control group (Placebo Comparator): Phase 1：50g glucose powder, dissolved in 250 mL of water
  Phase 2：The dosage is calculated at 0.5 grams per kilogram of adult body weight (e.g., a 60-kilogram adult would need to take 30 grams). Participants should dissolve the test product in water and drink it on an empty stomach before their first meal each day, continuing for 12 weeks.
  Interventions: Dietary Supplement: control group
- Commercially available resistant starch (Active Comparator): The dosage is calculated at 0.5 grams per kilogram of adult body weight (e.g., a 60-kilogram adult would need to take 30 grams). Subjects should dissolve the test product in water and drink it on an empty stomach before their first meal of the day.
  Interventions: Dietary Supplement: Commercially available resistant starch

INTERVENTIONS:
Dietary Supplement: RT-90 resistant tapioca starch — Within 5 minutes, consume resistant starch containing 50 g of total carbohydrates (total product weight 57 g), dissolved in 250 mL of water, and perform an oral glucose tolerance test to monitor blood sugar changes. After the test, the two groups will switch and consume resistant starch or glucose powder again after at least 1 week.
  Arms: RT-90 resistant tapioca starch
Dietary Supplement: control group — The subjects were asked to take a 50 g glucose powder dissolved in 250 mL of water within 5 minutes to conduct an oral glucose tolerance test to monitor blood sugar changes. After the test, the subjects were asked to empty their stomachs at least 1 week after the test and then switch to take RT-90 resistant starch or glucose powder again.
  Arms: control group
Dietary Supplement: Commercially available resistant starch — The dosage is calculated at 0.5 grams per kilogram of adult body weight (e.g., a 60-kilogram adult would need to take 30 grams). Participants should dissolve the test product in water and drink it on an empty stomach before their first meal each day, continuing for 12 weeks.
  Arms: Commercially available resistant starch

SUMMARY:
This study aims to investigate the effects of RT-90 resistant cassava starch on glycemic control using a human dietary trial and to evaluate its potential as a prebiotic fiber supplement. This study will assess the efficacy of RT-90 resistant cassava starch in improving glycemic control, body composition, and gut microbiome in healthy individuals.

DETAILED DESCRIPTION:
This study consisted of two phases.

The first phase was conducted in a randomized, cross-controlled manner. Before entering the study, participants maintained a normal diet and lifestyle for three consecutive days. Afterward, they entered the study and underwent a resistant starch assessment until the end of the study. Forty participants were randomly divided into two groups: 20 in each of the Weidan resistant starch group and the glucose powder group. Weidan resistant starch consists of tapioca resistant starch and glucose powder. Both groups consumed the sample within 5 minutes and then underwent an oral glucose tolerance test (OGTT). The participants fasted for 8-12 hours the day before the test (water was permitted). Blood samples (1 mL each) were collected at 0, 30, 60, 90, 120, and 180 minutes to monitor blood glucose levels. After the study, the two groups consumed either Weidan resistant starch or 50 g of glucose powder, each containing 50 g of total carbohydrates (57 g total product weight), dissolved in 250 mL of water, within 5 minutes, at least one week after the study. Blood glucose levels were monitored. After the study, the two groups alternated and consumed Weidan resistant starch or glucose powder again, followed by an oral glucose tolerance test and body composition measurements using the Inbody270 body composition analyzer.

The second phase of the study was conducted in a randomized, double-blind, placebo-controlled manner. Prior to entering the study, participants maintained a normal diet and lifestyle for three consecutive days. Afterward, they entered the study and underwent resistant starch assessment until completion. 75 subjects were randomly divided into three groups: the Weidan resistant starch group, the commercial resistant starch group, and the placebo control group. The ingredients of Weidan resistant starch are cassava resistant starch; the ingredients of commercial resistant starch are wheat resistant starch; and the placebo control group are natural cassava starch. The dosage is calculated based on 0.5 grams per kilogram of adult body weight (for example, a 60-kilogram adult needs to take 30 grams). The subjects were required to dissolve the test product in water and drink it on an empty stomach before their first meal each day for 12 weeks. The evaluation items at each follow-up visit included: (1) general physical examination (mental state, sleep, appetite, gastrointestinal symptoms, blood pressure, pulse and respiratory rate), (2) body measurement and body composition analysis (weight, BMI, waist circumference, hip circumference, subcutaneous fat thickness, skeletal muscle weight, body fat percentage and total water weight), (3) routine blood and biochemical examination, including red blood cell and white blood cell count, hemoglobin, hematocrit, mean corpuscular volume and platelets, renal function (urea nitrogen, creatinine, uric acid), thyroid hormone, liver function (AST, ALT, γ-GT and albumin), blood lipids (triglycerides, total cholesterol, free fatty acids, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol), electrolyte balance (sodium, potassium, chloride, phosphorus, calcium) and fasting blood glucose (blood volume was 15 mL, must fast for at least 8 hours), (4) diet and activity records (including 24-hour diet review and weekly gastrointestinal function symptom records), (5) analysis of intestinal related indicators, including short-chain fatty acids (SCFA) and intestinal flora (NGS). Samples were collected and analyzed at week 0 and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-65 years.
* Healthy subjects (BMI between 18.5-24.9 kg/m² for women and men).
* Subjects must be able to maintain a stable diet (based on the Ministry of Health and Welfare's daily dietary guidelines, with a tolerance of ± 10-15%) and physical activity (based on the World Health Organization's recommendations of 150-300 minutes of moderate-intensity exercise per week, or equivalent physical activity, with a tolerance of ± 20%) during the trial period.
* Subjects must understand the trial procedures and potential risks and benefits described in the consent form and be able to sign the consent form.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Subjects with endocrine abnormalities, major organ disease, or mental illness (as determined by a physician).
* Subjects found to be intolerant to the test sample during the trial.
* Subjects who develop a disease or take medications or health supplements that could affect the results of the trial during the trial period. (e.g., hypoglycemic (lipid)-lowering medications, probiotics, high-dose dietary fiber supplements, fish oil, or supplements high in polyunsaturated fatty acids).
* Chronic gastrointestinal diseases (e.g., diverticular disease, irritable bowel syndrome, or other intestinal diseases that may cause constipation).
* Use of antibiotics within the past three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Trial Changes in Fasting Blood Glucose from Baseline to End of Trial (Glycemic Index Test Phase) | Week 0 and 2
  Fasting blood glucose levels were measured at baseline and at the completion of the glycemic index (GI) test phase to assess short-term glycemic response.
  Blood Volume: 1 cc/times
Phase 2 Changes from Baseline to End of Trial (Prebiotic Assessment) | Week 0 to12
  Fasting blood glucose levels will be measured at baseline and 12 weeks after prebiotic supplementation to assess long-term metabolic response.
  Blood Draw Volume: 15 mL/dose
Phase 2 Changes from Baseline to End of Trial (Prebiotic Assessment | Week 0 and Week 12
  Ftool samples will be collected at Week 0 and Week 12 to analyze gut microbiota diversity.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, South, Taiwan